CLINICAL TRIAL: NCT03030794
Title: Alleviating Headache and Pain in GWI With Neuronavigation Guided rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H160047
Record Dates: First submitted 2017-01-04; First posted 2017-01-25 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2018-08

CONDITIONS: Gulf War Syndrome; Headache
Keywords: Gulf War Illness; Headache; Muscle Pain; Joint Pain; TMS
MeSH Terms: conditions — Persian Gulf Syndrome; Headache; Myalgia; Arthralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repetitive TMS (Active Comparator): Subjects will receive the repetitive transcranial magnetic stimulation study procedure.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- No (blocked) repetitive TMS (Placebo Comparator): Subjects will not receive the repetitive transcranial magnetic stimulation study procedure by blocking the stimulation between the coil and the head, but the audiovisual conditions will be mimicked.
  Interventions: Device: Repetitive transcranial magnetic stimulation (sham)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — A non-invasive method of brain stimulation that emits a magnetic pulse.
  Arms: Repetitive TMS
Device: Repetitive transcranial magnetic stimulation (sham) — No brain stimulation will be administered.
  Arms: No (blocked) repetitive TMS

SUMMARY:
This study aims to assess the effect of repetitive transcranial magnetic stimulation (rTMS) on Gulf War illness related headaches and pain.

DETAILED DESCRIPTION:
Headaches (HA) and wide spread pain are some of the most common debilitating symptoms in Gulf War Veterans (GWV) with Gulf War Illness (GWI). Migraine like HA and diffuse body pain were detected in 64% of GWV with GWI. This high prevalence of chronic HA and diffuse body pain conditions are often associated with neuropsychological dysfunction in mood, attention, memory and other systemic symptoms, which cast a profound negative impact on patients' quality of life. Unfortunately, conventional pharmacological treatments for GWI related headaches and pain (GWI-HAP) has not been shown to be effective and drugs such as narcotics contain many long term untoward psychosomatic and abusive side effects. Therefore, developing and validating non-invasive and low risk innovative treatment for this patient population is warranted. Transcranial Magnetic Stimulation (TMS) is currently a US FDA approved treatment for major depression and migraine HA.

ELIGIBILITY:
Criteria for veterans with Gulf War Illness headaches and pain:

Inclusion Criteria:

* Male or female between ages 18-65
* CDC Criteria for GWI
* Kansas Criteria for GWI
* International Headache Society Criteria for Migraine HA w/o aura
* Average Headache Exacerbation Intensity >3 on 0-10 NPRS
* Average Overall Daily Muscle Pain Intensity >3 on 0-10 NPRS
* Average Overall Daily Extremities Joint Pain Intensity >3 on 0-10 NPRS
* Headache Exacerbation/Attack ≥ 3 times/week, lasting >4 hrs in past 3 months

Exclusion Criteria:

* Pregnancy
* History of pacemaker implant
* Any ferromagnetic (e.g. bullet fragment, shrapnel, device implant) in the brain or body that will prohibit the patients from having a brain MRI
* History of dementia, major psychiatric diseases, or life threatening diseases
* Presence of any other chronic neuropathic pain states such as Complex Regional Pain Syndrome or Painful Peripheral Neuropathy
* History of seizure
* Pending litigation
* Low back pain with mechanical origins such as lumbar radiculopathy or radiculitis or lumbar facet arthropathy
* Lack of ability to understand the experimental protocol and to adequately communicate in English
* History of Traumatic Brain injury
* Chronic Tension or Cluster Headache
* Ongoing Cognitive Rehabilitation or Treatment of PTSD

Criteria for healthy veterans without Gulf War Illness headaches and pain:

Inclusion Criteria:

* Male or female between ages 18-65
* Served at least 30 consecutive days in the Persian Gulf between 8/90-7/91

Exclusion Criteria:

* CDC Criteria for GWI
* Kansas Criteria for GWI
* International Headache Society Criteria for Migraine HA w/o aura
* Average Headache Exacerbation Intensity >3 on 0-10 NPRS
* Average Overall Daily Muscle Pain Intensity >3 on 0-10 NPRS
* Average Overall Daily Extremities Joint Pain Intensity >3 on 0-10 NPRS
* Headache Exacerbation/Attack ≥ 3 times/week, lasting >4 hrs in past 3 months
* Pregnancy
* History of pacemaker implant
* Any ferromagnetic (e.g. bullet fragment, shrapnel, device implant) in the brain or body that will prohibit the patients from having a brain MRI
* History of dementia, major psychiatric diseases, or life threatening diseases
* Presence of any other chronic neuropathic pain states such as Complex Regional Pain Syndrome or Painful Peripheral Neuropathy
* History of seizure
* Pending litigation
* Low back pain with mechanical origins such as lumbar radiculopathy or radiculitis or lumbar facet arthropathy
* Lack of ability to understand the experimental protocol and to adequately communicate in English
* History of Traumatic Brain injury
* Chronic Tension or Cluster Headache
* Ongoing Cognitive Rehabilitation or Treatment of PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Daily Headache and Pain Log | 2 months for each subject (11 visits)
  This is a daily self-reporting log that tracks headache, muscle pain, and joint pain levels. The pain levels are scored from 0-10 with 10 being the worst possible pain.
Headache Impact Test 6 (HIT-6) | 2 months for each subject (11 visits)
  This 6-question form assesses the severity of headache pain and is scored with a range of 36-78. The higher score, the higher the impact of headaches on functional ability.
2 months for each subject (11 visits) | 2 months for each subject (11 visits)
  This assessment has 9 questions about pain level, relief, and interference. Pain level and interference questions range from 0-10, with 10 being the worst. Level of relief has a range of 0-100%, with 100% being complete relief.
Opioid Medication Assessment | 2 months for each subject (11 visits)
  This is a self-reporting log that tracks opioid medication usage. Average daily dosages are converted to equal-potent oral Morphine Sulfate dosage and reported in milligrams.
Mechanical-Visual Analogue Scale | 2 months for each subject (11 visits)
  This scale measures the level of headache, muscle, and joint pain at each visit. This ranges from 0-100, with 100 being the worst possible pain.

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | 2 months for each subject (11 visits)
  This is a 22-question self-report assessment that tracks symptoms over time. Each question ranges from 0-4, with 4 being very severe. The total NSI score ranges from 0-88.
Short-Form McGill Pain Questionnaire (SF-MPQ) | 2 months for each subject (11 visits)
  This self-reporting survey contains 15 questions that describe the type of pain. Each descriptor is scored between 0-3, with 3 being severe pain. The total score then ranges from 0-45. This questionnaire is filled out one each for joint pain and one for muscle pain.
New Clinical Fibromyalgia Diagnostic Criteria | 2 months for each subject (11 visits)
  This form contains a checklist of 19 possible areas for muscle pain. The checkmarks are tallied to give the Widespread Pain Index score, which ranges from 0-19. A score of 19 would suggest muscle pain in all 19 possible locations.
Revised Fibromyalgia Impact Questionnaire (FIQR) | 2 months for each subject (11 visits)
  This 3-part questionnaire measures the level of interference the pain causes, the overall impact of the pain, and intensity of the symptoms. There are a total of 21 questions, each with a range of 0-10, with 10 being either "very difficult" or "always." The FIQR total has a range of 0-210.
Conners Continuous Performance Test 2 (CPT2) | 2 months for each subject (11 visits)
  This is a 15-minute attention task administered on a laptop. The subject is prompted to press the spacebar as quickly as possible after every letter that appears on the screen except for the letter X. The exam is automatically scored by the program and reports omission rate and response latency. The attentional cognitive function is tracked by their change in these scores over time.
Hopkins Verbal Learning Test (HVLT) | 2 months for each subject (11 visits)
  This is a memory and recall task that requires the subject to memorize a list of 10 words and recall them. There are 3 trials and they are scored just by the number of words that can be recalled each time, which can be from 0-10 for a total range of 0-30 words. The second part of this test rates their recognition discrimination index by asking if certain words were on the original list. This is scored by taking the number of true positives and subtracting the false positives. The range for this is from 0-12, with 12 indicative of better discrimination within memory.
Trailmaking Test A&B | 2 months for each subject (11 visits)
  This is a timed test that is administered to assess executive function. Both tests have a series of numbers or numbers and letters that are to be connected in sequential order. The faster the completion time, the better the executive function.
This is a timed test that is administered to assess executive function. Both tests have a series of numbers or numbers and letters that are to be connected in sequential order. The faster the completion time, the better the executive function. | 2 months for each subject (11 visits)
  This is an administered IQ test that is designed to measure intelligence and cognitive ability in adults and older adolescents. There are several parts to the test, with each response being scored from 0-2 or 0-4 based on the quality of the answer or the completion time. The raw scores are then converted to scaled scores and summed to give the Full Scale score. The higher the Full Scale score, the higher the IQ classification.
Hamilton Rating Scale for Depression | 2 months for each subject (11 visits)
  This questionnaire rates the severity of depression in 21 questions. Each question either ranges from 0-2 or 0-4. The sum of the scores would give the total score, where a higher score would mean more severe depression.
36-Item Short Form Survey Instrument (SF-36) | 2 months for each subject (11 visits)
  This is a 38-question survey that assesses physical function, physical health limitations, emotional problem limitations, fatigue, emotional well-being, social functioning, pain, and general health. The scoring follows the official guidelines by RAND, where certain questions determine each health aspect. The questions are rated from 1-5, and then scored from 0-100. Each health aspect will have a range of 0-100, with 100 suggesting a more favorable health state.
Sleep Quality Assessment (PSQI) | 2 months for each subject (11 visits)
  This is self-reporting survey has 9 questions and determines the quality and patterns of sleep. Questions are either free-response or have a range from 0-3, with 3 being "more frequent" or "very bad." The responses will be scored based on the guidelines at the bottom of the page. The global PSQI score then has a range of 0-21, with 21 indicative of poor sleep quality.
Insomnia Severity Index | 2 months for each subject (11 visits)
  This survey has 7 questions that rate the severity of insomnia problems. All questions range from 0-4 and the sum of the answers would give the total score. The total score range from 0-28, with 28 being severe clinical insomnia.
Flinders Fatigue Scale | 2 months for each subject (11 visits)
  This questionnaire contains 7 questions in order to determine the level of fatigue one is experiencing. The questions range from 1-5, with 5 being "extremely" or "entirely." The higher one scores, the more severe the fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Leung, M.D., Principal Investigator — VA San Diego Health Care System
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Veteran Affairs Hospital, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung A, Donohue M, Xu R, Lee R, Lefaucheur JP, Khedr EM, Saitoh Y, Andre-Obadia N, Rollnik J, Wallace M, Chen R. rTMS for suppressing neuropathic pain: a meta-analysis. J Pain. 2009 Dec;10(12):1205-16. doi: 10.1016/j.jpain.2009.03.010. Epub 2009 May 23. PMID 19464959
- [Background] Leung A, Shukla S, Fallah A, Song D, Lin L, Golshan S, Tsai A, Jak A, Polston G, Lee R. Repetitive Transcranial Magnetic Stimulation in Managing Mild Traumatic Brain Injury-Related Headaches. Neuromodulation. 2016 Feb;19(2):133-41. doi: 10.1111/ner.12364. Epub 2015 Nov 10. PMID 26555886
- [Derived] Lei K, Kunnel A, Metzger-Smith V, Golshan S, Javors J, Wei J, Lee R, Vaninetti M, Rutledge T, Leung A. Diminished corticomotor excitability in Gulf War Illness related chronic pain symptoms; evidence from TMS study. Sci Rep. 2020 Oct 28;10(1):18520. doi: 10.1038/s41598-020-75006-8. PMID 33116195